CLINICAL TRIAL: NCT05950139
Title: Pilot Study of a Prophylactic Cancer Peptide Vaccine in Advanced ALK+ NSCLC
Brief Title: Peptide Vaccine To Prevent Acquired Resistance In Patients With Advanced ALK+ NSCLC
Acronym: ARCHER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Oncovir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J23120; IRB00398546 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: NSCLC Stage IV; ALK Fusion Protein Expression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Protein Subunit Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Advanced ALK+ NSCLC (Experimental): All patients will receive the intervention
  Interventions: Biological: Peptide vaccine

INTERVENTIONS:
Biological: Peptide vaccine — Peptide vaccine

SUMMARY:
The purpose of this study is to evaluate the safety of a cancer peptide vaccine to prevent or delay acquired resistance in advanced ALK+ lung cancer patients currently on ALK targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of stage IV NSCLC (or recurrent NSCLC not a candidate for definitive multimodality therapy)
2. Documented ALK rearrangement as detected by: (1) fluorescence in situ hybridization (FISH), (2) immuno-histochemistry (IHC), (3) tissue next-generation sequencing (NGS), or (4) circulating tumor DNA (ctDNA) NGS
3. Ongoing treatment with crizotinib, ceritinib, alectinib, brigatinib, or lorlatinib with at least stable disease ≥ 4 months
4. No known presence of the specific ALK acquired resistance alterations targeted by the study vaccine
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
6. Males or females at least 18 years old

Exclusion Criteria:

1. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Adequately resected non-melanoma skin cancer, curatively treated in-situ disease, and other solid tumors treated with potentially curative therapy are allowed.
2. Cytotoxic chemotherapy within 14 days of first dose of study vaccine or concurrent with study vaccine
3. Anti-neoplastic immunotherapy within 28 days of first dose of study vaccine or concurrent with study vaccine
4. Systemic immune suppression:

   1. Use of chronic oral or systemic steroid medication (topical or inhalational steroids are permitted)
   2. Other clinically relevant systemic immune suppression
5. Symptomatic central nervous system (CNS) metastasis. Asymptomatic CNS disease requiring increasing dose of corticosteroids within 7 days prior to study enrollment is also not permitted
6. Current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Patients with leptomeningeal disease and without cord compression are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 2 years
  The safety of administering the ALK peptide vaccine will be assessed by the occurrence of the following adverse events:
  * Grade 3 or above drug-related toxicities
  * Drug-related toxicity by grade
  * Vaccine site reactions after vaccine injections
  * Immune-related adverse events (AEs)
  * Unacceptable toxicities
  * Treatment-emergent changes from normal to abnormal values in key laboratory parameters
Vaccine-specific immune response | Up to 2 years
  Vaccine-specific response will be evaluated by the fold change in interferon-producing mutant-ALK-specific CD8 and CD4 T cells in the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Lam, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States